CLINICAL TRIAL: NCT05762055
Title: Prospective Comparative Analysis Evaluating Radiographic and Clinical Outcomes of Stand-Alone Anterior Cervical Discectomy and Fusion Interbody Cages With nanoLOCK Osseointegrative Technology
Brief Title: Prospective Comparative Analysis of ACDF vs Fusion Interbody Cages With nanoLOCK Osseointegrative Technology
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Salah Aoun, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-1092
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cervical Radiculopathy; Cervical Myelopathy
Keywords: spine; cervical; discectomy; bony fusion; dysphagia; radiographic fusion; radiographic adjacent segment disease
MeSH Terms: conditions — Radiculopathy; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Medtronic Titan Endoskeleton TCS zero-profile, stand-alone interbody cages with nanoLOCK osseointegrative technology will be implanted for participants in this group
  Interventions: Device: Titan nanoLOCK interbody cage
- Control Group (Experimental): Participants in this arm will receive an alternative interbody cage system that does not employ nanoLOCK ossteointegrative technology.
  Interventions: Device: ACDF interbody cage

INTERVENTIONS:
Device: Titan nanoLOCK interbody cage — Medtronic Titan Endoskeleton TCS zero-profile, stand-alone interbody cages with nanoLOCK osseointegrative technology
  Other Names: Titan nanoLOCK®
  Arms: Intervention Group
Device: ACDF interbody cage — Anterior cervical discectomy and fusion (ACDF) is an alternative interbody cage system that does not employ nanoLOCK ossteointegrative technology
  Arms: Control Group

SUMMARY:
Study team will plan a prospective, randomized control trial using our institution's spine clinical outcomes registry. Eligible patients undergoing ACDF (see inclusion criteria listed below) will be randomized to an Intervention or Control Group, which will differ according to the interbody cage used during the procedure. In the Intervention Group (100 patients), Medtronic Titan Endoskeleton TCS zero-profile, stand-alone interbody cages with nanoLOCK osseointegrative technology will be implanted at each treated level. In the Control Group (100 patients), patients will receive an alternative interbody cage system that does not employ nanoLOCK ossteointegrative technology. Interbody cages used in the Control Group (along with the decision to apply anterior plate fixation) will be determined according to surgeon preference. There will be no blinding to the type of implant used. Standard demographic and procedural variables will be collected for all patients (including history of diabetes, tobacco, use, prior use of oral corticosteroids, number of levels fused, and presence of bicortical screw placement). Clinical and radiographic outcomes in the Intervention and Control Groups will be directly compared.

DETAILED DESCRIPTION:
Aim 1: Examine the effect of nanoLOCK technology on rates of postoperative dysphagia after ACDF.

Aim 2: Evaluate the effect of nanoLOCK technology on radiographic fusion.

Aim 3: Evaluate how nanoLOCK technology influences the development of radiographic adjacent segment disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* Subjects undergoing ACDF surgery for degenerative pathology (one, two or three levels)
* Subjects with no prior history of cervical spine surgery
* Subjects with complete/usable data

Exclusion Criteria:

* Subjects under the age of 18
* Subjects not undergoing ACDF surgery
* Subjects with prior cervical spine surgery
* Subjects with cervical neoplastic or infectious disease pathology
* Subjects with cervical trauma pathology
* ACDF performed at C2-3
* Subjects with incomplete/unusable data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patient reported dysphagia events measured by Eat-10 assessment tool | Postoperative at Day 1
  Number of patient reported dysphagia events (incidence & severity ) is measured by Eating Assessment Tool (EAT-10) post surgery at day1 which is self-administered, symptom-specific outcome instrument for dysphagia. It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem.
Number of patient reported dysphagia events measured by Eat-10 assessment tool | 2 weeks following surgery
  Number of patient reported dysphagia events (incidence & severity ) is measured by Eating Assessment Tool (EAT-10) post surgery at day1 which is self-administered, symptom-specific outcome instrument for dysphagia. It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem.
Number of patient reported dysphagia events measured by Eat-10 assessment tool | 3 months following surgery
  Number of patient reported dysphagia events (incidence & severity ) is measured by Eating Assessment Tool (EAT-10) post surgery at day1 which is self-administered, symptom-specific outcome instrument for dysphagia. It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem.
Number of patient reported dysphagia events measured by Eat-10 assessment tool | 6 months following surgery
  Number of patient reported dysphagia events (incidence & severity ) is measured by Eating Assessment Tool (EAT-10) post surgery at day1 which is self-administered, symptom-specific outcome instrument for dysphagia. It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem.
Number of patient reported dysphagia events measured by Eat-10 assessment tool | 12 months following surgery
  Number of patient reported dysphagia events (incidence & severity ) is measured by Eating Assessment Tool (EAT-10) post surgery at day1 which is self-administered, symptom-specific outcome instrument for dysphagia. It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem.
Dysphagia as measured by SWAL-QOL assessment tool | Postoperative at day 1
  Dysphagia is measured by SWAL-QOL assessment tool which is designed to find out how one's swallowing problem has been affecting their day-to-day quality of life. Scoring in each domain is calculated by the sums of scores for each item expressed as a percentage of the maximum possible domain score. A total SWAL-QOL score is derived by summing each domain score and dividing by 10 giving a total SWAL-QOL score that ranges between 0 and 100 (worst-best).
Dysphagia as measured by SWAL-QOL assessment tool | 2 weeks following surgery
  Dysphagia is measured by SWAL-QOL assessment tool which is designed to find out how one's swallowing problem has been affecting their day-to-day quality of life. Scoring in each domain is calculated by the sums of scores for each item expressed as a percentage of the maximum possible domain score. A total SWAL-QOL score is derived by summing each domain score and dividing by 10 giving a total SWAL-QOL score that ranges between 0 and 100 (worst-best).
Dysphagia as measured by SWAL-QOL assessment tool | 3 months following surgery
  Dysphagia is measured by SWAL-QOL assessment tool which is used in understanding quality of life in swallowing disorders. Scoring in each domain is calculated by the sums of scores for each item expressed as a percentage of the maximum possible domain score. A total SWAL-QOL score is derived by summing each domain score and dividing by 10 giving a total SWAL-QOL score that ranges between 0 and 100 (worst-best).
Dysphagia as measured by SWAL-QOL assessment tool | 6 months following surgery
  Dysphagia is measured by SWAL-QOL assessment tool which is designed to find out how one's swallowing problem has been affecting their day-to-day quality of life. Scoring in each domain is calculated by the sums of scores for each item expressed as a percentage of the maximum possible domain score. A total SWAL-QOL score is derived by summing each domain score and dividing by 10 giving a total SWAL-QOL score that ranges between 0 and 100 (worst-best).
Dysphagia as measured by SWAL-QOL assessment tool | 12 months following surgery
  Dysphagia is measured by SWAL-QOL assessment tool which is designed to find out how one's swallowing problem has been affecting their day-to-day quality of life. Scoring in each domain is calculated by the sums of scores for each item expressed as a percentage of the maximum possible domain score. A total SWAL-QOL score is derived by summing each domain score and dividing by 10 giving a total SWAL-QOL score that ranges between 0 and 100 (worst-best).
Degree of radiographic fusion | 6 weeks following surgery
  Degree of radiographic fusion is measured by quantifying (count of) the presence of bony trabeculae crossing the interface between the implant and adjacent levels as obtained via CT of the cervical spine.
Degree of radiographic fusion | 3 months following surgery
  Degree of radiographic fusion is measured by quantifying (count of) the presence of bony trabeculae crossing the interface between the implant and adjacent levels as obtained via CT of the cervical spine.
Degree of radiographic fusion | 6 months following surgery
  Degree of radiographic fusion is measured by quantifying (count of) the presence of bony trabeculae crossing the interface between the implant and adjacent levels as obtained via CT of the cervical spine.
Degree of radiographic fusion | 12 months following surgery
  Degree of radiographic fusion is measured by quantifying (count of) the presence of bony trabeculae crossing the interface between the implant and adjacent levels as obtained via CT of the cervical spine.
Incidence of radiographic adjacent segment disease | 6 months following surgery
  Incidence of radiographic adjacent segment disease is measured by quantifying (number of occurrence) the following parameters (i.e., Suprajacent and/or subjacent level kyphosis; Vacuum disc phenomenon at adjacent level discs; Adjacent level compression deformity) on postoperative imaging
Incidence of radiographic adjacent segment disease | 12 months following surgery
  Incidence of radiographic adjacent segment disease is measured by quantifying (number of occurrence) the following parameters (i.e., Suprajacent and/or subjacent level kyphosis; Vacuum disc phenomenon at adjacent level discs; Adjacent level compression deformity) on postoperative imaging

SECONDARY OUTCOMES:
Percentage of participants experiencing neck pain | Baseline (Pre-op)
  Percentage of participants experiencing neck pain is assessed using VAS-neck questionnaire. Possible scores range from 0-10, where 0=no pain and 10= worst pain imaginable.
Percentage of participants experiencing neck pain | 6 weeks following surgery
  Percentage of participants experiencing neck pain is assessed using Vissual Analogue Scale (VAS)-neck questionnaire. Possible scores range from 0-10, where 0=no pain and 10= worst pain imaginable.
Percentage of participants experiencing neck pain | 3 months following surgery
  Percentage of participants experiencing neck pain is assessed using VAS-neck questionnaire. Possible scores range from 0-10, where 0=no pain and 10= worst pain imaginable.
Percentage of participants experiencing neck pain | 6 months following surgery
  Percentage of participants experiencing neck pain is assessed using VAS-neck questionnaire. Possible scores range from 0-10, where 0=no pain and 10= worst pain imaginable.
Percentage of participants experiencing neck pain | 12 months following surgery
  Percentage of participants experiencing neck pain is assessed using VAS-neck questionnaire. Possible scores range from 0-10, where 0=no pain and 10= worst pain imaginable.
Percentage of participants showing functional improvement | Baseline (Pre-op)
  Percentage of participants showing functional improvement is assessed using Neck Disability Index (NDI) questionnaire. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.
Percentage of participants showing functional improvement | 6 weeks following surgery
  Percentage of participants showing functional improvement is assessed using Neck Disability Index (NDI) questionnaire. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.
Percentage of participants showing functional improvement | 3 months following surgery
  Percentage of participants showing functional improvement is assessed using Neck Disability Index (NDI) questionnaire. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.
Percentage of participants showing functional improvement | 6 months following surgery
  Percentage of participants showing functional improvement is assessed using Neck Disability Index (NDI) questionnaire. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.
Percentage of participants showing functional improvement | 12 months following surgery
  Percentage of participants showing functional improvement is assessed using Neck Disability Index (NDI) questionnaire. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.
Number of participants who experienced overall complications | 3 years following surgery
  Overall complication rate is measured by number of participants who experienced overall complications (including instrumentation fracture, cage subsidence, revision surgery, and wound breakdown/infection)
Percentage of participants reporting functional outcomes as measured by PROMIS-29 | Baseline (Pre-op)
  Percentage of participants reporting functional outcomes is measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire which contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 NRS. The raw score of each domain is converted into a standardized score with a mean of 50 and a SD of 10 for the general population in the US (T-Score).
Percentage of participants reporting functional outcomes as measured by PROMIS-29 | 6 weeks following surgery
  Percentage of participants reporting functional outcomes is measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire which contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 NRS. The raw score of each domain is converted into a standardized score with a mean of 50 and a SD of 10 for the general population in the US (T-Score).
Percentage of participants reporting functional outcomes as measured by PROMIS-29 | 3 months following surgery
  Percentage of participants reporting functional outcomes is measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire which contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 NRS. The raw score of each domain is converted into a standardized score with a mean of 50 and a SD of 10 for the general population in the US (T-Score).
Percentage of participants reporting functional outcomes as measured by PROMIS-29 | 6 months following surgery
  Percentage of participants reporting functional outcomes is measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire which contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 NRS. The raw score of each domain is converted into a standardized score with a mean of 50 and a SD of 10 for the general population in the US (T-Score).
Percentage of participants reporting functional outcomes as measured by PROMIS-29 | 12 months following surgery
  Percentage of participants reporting functional outcomes is measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire which contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 NRS. The raw score of each domain is converted into a standardized score with a mean of 50 and a SD of 10 for the general population in the US (T-Score).

CONTACTS AND LOCATIONS:
Overall Officials: Salah Aoun, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No